CLINICAL TRIAL: NCT03183050
Title: MEND 2: Making Treatment Decisions Using Genomic Testing
Acronym: MEND2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other); Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Suzanne C. O'Neill, Associate Professor, Georgetown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-1117
Record Dates: First submitted 2017-06-05; First posted 2017-06-09 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Question Prompt List (Experimental): Paper booklet including question prompt list.
  Interventions: Behavioral: Question Prompt List

INTERVENTIONS:
Behavioral: Question Prompt List — Patients receive a booklet that contains questions regarding their diagnosis, testing and treatment.

SUMMARY:
Clinical guidelines for women with early stage breast cancer integrate genomic tumor profiling tests such as the Oncotype DX Recurrence Score to refine recurrence estimates and systemic therapy selection when combined with existing markers. Guidelines suggest that the 25% with a high Score benefit from chemotherapy and the 50% with a low Score can safely avoid chemotherapy. Many challenges remain to maximize the benefits of testing prior to release of trial results in the next year. Strong clinical communication can impact proximal outcomes of patient comprehension, treatment preferences and satisfaction, involvement in care decisions as well as longer-term outcomes of treatment adherence and QOL. These proximal outcomes can be influenced by patient activation interventions utilizing a question prompt list (QPL). In the context of patients receiving Oncotype DX testing, the QPL could allow them to better understand the rationale for their oncologist's treatment recommendation, what it means for managing their disease, and encourage alignment of treatment preferences and selection with the Recurrence Score. Research is conducted in two phases to test the feasibility and impact of the QPL. In Phase 1, the draft QPL will be revised based on in-depth interviews with patients (N=20) and medical oncologists (N=10). Phase 2 will be a single-arm trial (N=75) to demonstrate feasibility and preliminarily assess the impact of the QPL on key outcomes.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer among US women, with more than 230,000 new diagnoses and 40,000 deaths each year, along with decrements in quality of life. Half of all newly-diagnosed patients are affected with estrogen-receptor positive, early-stage disease. Clinical guidelines for these women integrate genomic tumor profiling tests such as the Oncotype DX® Recurrence Score to refine recurrence estimates and systemic therapy selection when combined with existing markers. Thousands of women receive testing each year. While these women should all receive hormonal therapy, guidelines suggest that the 25% with a high Score benefit from additional chemotherapy and the 50% with a low Score can safely avoid chemotherapy. Appropriate treatment for the 25% of women with intermediate Recurrence Scores remains unclear until clinical trial (TAILORx) results are released in the next year.

Despite continuing dissemination, many challenges remain to maximize the benefits offered by testing and refined treatment selection. TAILORx results will continue to strengthen the evidence for clinical utility and increase testing rates. An effective intervention should be ready to respond to this increasing need. Communication can influence more proximal outcomes, including patient comprehension of their disease and its treatments, treatment preferences and satisfaction, involvement in care decisions as well as longer-term outcomes of treatment adherence and quality of life. This trial will test the feasibility and impact of a patient activation intervention to support effective integration of the Recurrence Score into clinical encounters and treatment decisions. Patient activation interventions utilizing a question prompt list (QPL) can impact proximal outcomes of preferences, comprehension, satisfaction and involvement. Women with newly-diagnosed breast cancer will be recruited to a single-arm trial to demonstrate feasibility and preliminarily assess the impact of the QPL on key outcomes. Aims are to:

Aim 1. Examine intervention feasibility. Feasibility will be examined in 3 areas: 1) patient and oncologist acceptability, 2) participant recruitment and retention, and 3) intervention dosage and fidelity.

Aim 2. Evaluate intervention effects on comprehension and treatment preferences. 2a: Participants will demonstrate significant increases in comprehension about their disease and its treatments from pre- to post-QPL. 2b: Participants will be more likely to report Score-concordant preferences from pre to post-QPL.

Aim 3. Assess potential intervention mechanisms on comprehension, preferences and satisfaction. 3a: Patient comprehension and satisfaction will be higher following encounters with greater shared decision making, greater perceived communication quality, and more frequent discussion of risks/benefits of treatments. 3b: Patient preferences will likely be more Score-concordant following encounters with greater shared decision making, greater perceived communication quality, and more frequent discussion of risks/benefits of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40-75 who receive Oncotype DX testing are eligible.

Exclusion Criteria:

* Cognitive impairment that precludes informed consent and inability to converse in English given the focus on communication in this study. Clinical communication between providers and patients with limited English proficiency is beyond the scope of this work.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne C O'Neill, PhD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Medstar Cancer Network, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Yes
Data will include self-reported survey data, data obtained from chart review and audio recorded encounters. We will make de-identified data available by request to investigators not associated with the study. Priority for sharing of data will be given to junior faculty and/or faculty interested in questions related to translational science. Any requests for data from non-study investigators will be reviewed by the investigative team to ensure that it does not conflict with planned analyses, is otherwise respectful of the study participants, and complies with all relevant IRB and HIPAA regulations.
Supporting Information: Study Protocol
Time Frame: Clean, de-identified dataset can be made available once analyses associated with study aims are complete.
Access Criteria: Investigator must be willing to follow all procedures requested by IRB of record.

REFERENCES:
- [Result] O'Neill SC, Vadaparampil ST, Street RL Jr, Moore TF, Isaacs C, Han HS, Augusto B, Garcia J, Lopez K, Brilleman M, Jayasekera J, Eggly S. Characterizing patient-oncologist communication in genomic tumor testing: The 21-gene recurrence score as an exemplar. Patient Educ Couns. 2021 Feb;104(2):250-256. doi: 10.1016/j.pec.2020.08.037. Epub 2020 Sep 3. PMID 32900604
- [Result] Jayasekera J, Vadaparampil ST, Eggly S, Street RL Jr, Foster Moore T, Isaacs C, Han HS, Augusto B, Garcia J, Lopez K, O'Neill SC. Question Prompt List to Support Patient-Provider Communication in the Use of the 21-Gene Recurrence Test: Feasibility, Acceptability, and Outcomes. JCO Oncol Pract. 2020 Oct;16(10):e1085-e1097. doi: 10.1200/JOP.19.00661. Epub 2020 May 28. PMID 32463763

RESULTS

PARTICIPANT FLOW:
Groups:
- Received QPL: Each participant of this single-arm trial received the QPL
Period: Overall Study
Arm/Group | Received QPL
Started | 88
Completed | 65
Not Completed | 23
Not completed — Lost to Follow-up | 23

BASELINE CHARACTERISTICS:
Population: A total of 88 patients consented to the trial, but only 65 patients completed final screening and baseline interview.
Arm/Group | Received QPL
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 53
  More than one race | 0
  Unknown or Not Reported | 1
Knowledge Related to Testing and Treatment [Mean (Standard Deviation); unit: units on a scale] — Knowledge was measured for testing, treatment and overall. Responses included true/false/don't know with a point per correct answer. Testing knowledge was assessed with a 12-item scale from Richman et al. (2011), with an overall score from 0-12. Treatment knowledge was assessed with 5 items from the Breast Cancer Systemic Therapy Decision Quality Instrument (Lee et al., 2014; overall score of 0-5). Knowledge was scored separately for testing and treatment, as well as summed for a total knowledge score (0-17), which is used as the primary outcome. Higher scores correspond to more knowledge.
  units on a scale | 10.95 (2.98)

OUTCOME MEASURES:

1. Primary Outcome: Knowledge Related to Testing and Treatment
Description: Knowledge was measured for testing, treatment and overall. Responses included true/false/don't know with a point per correct answer. Testing knowledge was assessed with a 12-item scale from Richman et al. (2011), with an overall score from 0-12. Treatment knowledge was assessed with 5 items from the Breast Cancer Systemic Therapy Decision Quality Instrument (Lee et al., 2014; overall score of 0-5). Knowledge was scored separately for testing and treatment, as well as summed for a total knowledge score (0-17), which is used as the primary outcome. Higher scores correspond to more knowledge.
Time Frame: One month
Population: All consented participants who completed both time points
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Received QPL
Number analyzed (Participants) | 65
units on a scale | 12.36 (13.0)

ADVERSE EVENTS:
Time Frame: Participants were able to report adverse events at any time during their participation, approximately three months from consent to completion of all study activities.
Arm/Group | Received QPL
All-Cause Mortality (participants affected / at risk) | 0/88
Serious Adverse Events (participants affected / at risk) | 0/88
Other Adverse Events (participants affected / at risk) | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT03183050/Prot_SAP_000.pdf